CLINICAL TRIAL: NCT03526978
Title: A Randomized, Double-blind, Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of Sabin Inactivated Poliovirus Vaccine (Vero Cell) in 2-month-old Infants
Brief Title: An Immunogenicity and Safety Study of Sabin Inactivated Poliovirus Vaccine (Vero Cell) in 2-month-old Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-sIPV-3001
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Poliomyelitis
Keywords: Sabin strain; Inactivated poliovirus vaccine; poliomyelitis; safety; immunogenicity; infant
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The investigational vaccine was manufactured by Sinovac Vaccine Technology Co., Ltd.
  Intervention: investigational sIPV
  Interventions: Biological: Investigational sIPV
- Control Group (Active Comparator): The control vaccine was manufactured by Sanofi Pasteur Company. Intervention: control IPV
  Interventions: Biological: Control IPV

INTERVENTIONS:
Biological: Investigational sIPV — Three intramuscular injections of the investigational vaccine (0.5 ml) on Day 0, Day 30 and Day 60 respectively; Single intramuscular injection of the investigational vaccine (0.5 ml) at 18 months; Intervention: investigational sIPV
  Arms: Experimental Group
Biological: Control IPV — Three intramuscular injections of the control vaccine (0.5 ml) on Day 0, Day 30 and Day 60 respectively; Single intramuscular injection of the control vaccine (0.5 ml) at 18 months; Intervention:control IPV
  Arms: Control Group

SUMMARY:
The purpose of this phase III study is to evaluate the immunogenicity and safety of Sabin Inactivated Poliovirus Vaccine (Vero cell) in 2-month-old infants.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, controlled randomized, double-blind, controlled clinical trial clinical trial. The purpose of this study is to evaluate the immunogenicity and safety of Sabin Inactivated Poliovirus Vaccine (Vero cell) manufactured by Sinovac Vaccine Technology Co., Ltd in 2-month-old infants. The control vaccine is a commercialized Inactivated Poliovirus Vaccine manufactured by Sanofi Pasteur company. 1200 healthy infants between 60-90 days will be randomly assigned into experimental group or control group in the ratio 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 60-90 days old;
* Healthy volunteers who fulfill all the required conditions for receiving the investigational vaccine as established by medical history and clinical examination and determined by investigators;
* Proven legal identity;
* Participants or guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrolment;
* Complying with the requirement of the study protocol;

Exclusion Criteria:

* Prior vaccination with Poliovirus Vaccine;
* History of allergy to any vaccine, or any ingredient of the vaccine, or serious adverse reaction(s) to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc;
* Congenital malformation, developmental disorders, genetic defects, or severe malnutrition;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* Severe nervous system disease (epilepsy, seizures or convulsions) or mental illness;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) prior to study entry;
* Blood product prior to study entry;
* Any other investigational medicine(s) within 30 days prior to study entry;
* Any live attenuated vaccine within 14 days prior to study entry;
* Any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Axillary temperature > 37.0 °C;
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators;

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCRs) of each group after primary immunization. | 90 days
  Subjects whose pre-immune antibody level < 1:8 and post-immune antibody level ≥ 1:8, or those whose pre-immune antibody level ≥ 1:8 and the increase of post-immune antibody level ≥ 4 folds are considered seroconverted. Primary vaccination schedule: 3 doses with one month interval between doses (i.e., month 0, 1, 2).

SECONDARY OUTCOMES:
The incidences of solicited adverse events (AEs) of each group. | 7 days
  Solicited AEs occurred within 7 days after each injection will be collected.
The incidences of unsolicited adverse events (AEs) of each group. | 30 days
  Unsolicited AEs occurred within 30 days after each injection will be collected.
The incidence of serious adverse events (SAEs) during the period of safety monitoring of each group. | 90-420 days.
  SAEs during the period of safety monitoring will be collected.
The post-immune antibody positive rate of each group after primary immunization. | 90 days
  Subjects whose post-immune antibody level ≥ 1:8 are considered antibody positive. Primary vaccination schedule: 3 doses with one month interval between doses (i.e., month 0, 1, 2).
The post-immune geometric mean titer (GMT) of each group after primary immunization. | 90 days.
  GMT of each group after primary immunization which lasts 60 days.
The geometric mean fold increase (GMI) of each group after primary immunization. | 90 days
  The GMI is the increase of post-immune GMT from pre-immune GMT.
The percentage of subjects with antibody ≥ 1:64 of each group after primary immunization. | 90 days
  Percentage of subjects with antibody ≥ 1:64 of each group after three-dose
The antibody positive rate of each group before booster dose. | 420 days
  Subjects whose post-immune antibody level ≥ 1:8 are considered antibody positive. A booster dose at the age of 18months.
The geometric mean titer (GMT) of each group before booster dose. | 420 days.
  GMT of each group before booster dose which occurred at the age of 18months.
The geometric mean fold increase (GMI) of each group before booster dose. | 420 days
  The GMI is the increase of post-immune GMT from pre-i mmune GMT.
The percentage of subjects with antibody ≥ 1:64 of each group before booster dose. | 420 days
  Percentage of subjects with antibody ≥ 1:64 of each group before booster dose which occurred at the age of 18months.
The post-immune antibody positive rate of each group after booster dose. | 570 days
  Subjects whose post-immune antibody level ≥ 1:8 are co
  nsidered antibody positive
The post-immune geometric mean titer (GMT) of each group after booster dose. | 570 days
  GMT of each group after booster dose. The booster dose at the age of 18months
The geometric mean fold increase (GMI) of each group after booster dose. | 570 days
  The GMI is the increase of post-immune GMT from pre-immune GMT.
The percentage of subjecs with antibody ≥ 1:64 of each group after booster dose. | 570 days
  Percentage of subjecs with antibody ≥ 1:64 of each group after booster dose which occurred at the age of 18months.

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Pizhou County Center for Disease Control and Prevention, Pizhou, Jiangsu, China

REFERENCES:
- [Derived] Hu Y, Wang J, Zeng G, Chu K, Jiang D, Zhu F, Ying Z, Chen L, Li C, Zhu F, Yin W. Immunogenicity and Safety of a Sabin Strain-Based Inactivated Polio Vaccine: A Phase 3 Clinical Trial. J Infect Dis. 2019 Oct 8;220(10):1551-1557. doi: 10.1093/infdis/jiy736. PMID 30958543